CLINICAL TRIAL: NCT05087381
Title: Randomized-controlled Trial of the Effectiveness of COVID-19 Early Treatment in Community With Fluvoxamine, Bromhexine, Cyproheptadine, and Niclosamide in Decreasing Recovery Time
Brief Title: Randomized-controlled Trial of the Effectiveness of COVID-19 Early Treatment in Community
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Department of Medical Services Ministry of Public Health of Thailand (Other Government); Ministry of Health, Thailand (Other Government); Mahidol University (Other); Ramathibodi Hospital (Other); QIMR Berghofer Medical Research Institute (Other); Yamagata Prefectural Central Hospital (Unknown); The University of Western Australia (Other); Mae Fah Luang University (Other); King Chulalongkorn Memorial Hospital (Other); Washington University School of Medicine (Other); Vibhavadi Hospital (Unknown); Thanyarak Pattani Hospital (Unknown)
Responsible Party: Principal Investigator, Dhammika Leshan Wannigama, MD, Fellow and Scientist, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 64197
Record Dates: First submitted 2021-10-19; First posted 2021-10-21 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Treatment Efficacy
Keywords: COVID-19; Coronavirus; Treatment; Viral shedding; Coronavirus Infections; Respiratory Tract Infections; Anti-Infective Agents; Fluvoxamine; Bromhexine; Cyproheptadine; Niclosamide; Pneumonia, Viral; Early treatment
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Tract Infections; Pneumonia, Viral | interventions — Fluvoxamine; Bromhexine; Cyproheptadine; Niclosamide

STUDY DESIGN:
Intervention Model Description: Open label, multiarm, prospective, randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Fluvoxamine Arm (Experimental): The subjects received fluvoxamine (immediate release) 50 mg, 1 tablet in the morning and 50 mg 2 tablets before bedtime, orally after meals. For a total of 14 days, the first two days and the last two days, 50 mg 1 tablet in the morning and 50 mg 1 tablet at bedtime.
  Interventions: Drug: FluvoxaMINE Maleate 50 MG
- Fluvoxamine in Combination with Bromhexine Arm (Experimental): The subjects received fluvoxamine (immediate release) 50 mg, 1 tablet in the morning and 50 mg 2 tablets before bedtime, orally after meals. For a total of 14 days, the first two days and the last two days, 50 mg 1 tablet in the morning and 50 mg 1 tablet at bedtime. Co- administration with bromhexine 8 mg, 1 tablet twice taken after meals and taken at least 8 hours apart, for 10 days.
  Interventions: Combination Product: Fluvoxamine, Bromhexine
- Fluvoxamine in Combination with Cyproheptadine Arm (Experimental): The subjects received fluvoxamine (immediate release) 50 mg, 1 tablet in the morning and 50 mg 2 tablets before bedtime, orally after meals. For a total of 14 days, the first two days and the last two days, 50 mg 1 tablet in the morning and 50 mg 1 tablet at bedtime. Co- administration with cyproheptadine 4 mg, 1 tablet, three times, orally after meals and should be taken every 8 hours apart, for 14 days.
  Interventions: Combination Product: Fluvoxamine, Cyproheptadine
- Niclosamide Arm (Experimental): The subjects received 1 tablet of niclosamide 1000 mg orally in divided doses twice a day. After meals in the morning and evening for a total of 14 days.
  Interventions: Drug: Niclosamide Pill
- Niclosamide in Combination with Bromhexine Arm (Experimental): The subjects received 1 tablet of niclosamide 1000 mg orally in divided doses twice a day. After meals in the morning and evening for a total of 14 days. Co-administration with bromhexine 8 mg, 1 tablet twice taken after meals and taken at least 8 hours apart, for 10 days.
  Interventions: Combination Product: Niclosamide, Bromhexine
- Usual Care Arm (No Intervention): The control group received treatment according to the latest usual care medical guidelines provide by ministry of Thailand at that time.

INTERVENTIONS:
Drug: FluvoxaMINE Maleate 50 MG — The subjects received fluvoxamine (immediate release) 50 mg, 1 tablet in the morning and 50 mg 2 tablets before bedtime, orally after meals. For a total of 14 days, the first two days and the last two days, 50 mg 1 tablet in the morning and 50 mg 1 tablet at bedtime.
  All enrolled patients will be provided a thermometer as well as a fingertip probe pulse oximeter, with the specific instructions to monitor both temperature at oxygen saturation at the time of daily oral administration of drug. In addition, Oropharyngeal swab samples will be collected for viral shedding as measured by PCR on days 0, 7 and 14. Fecal and blood samples will be collected for viral shedding as measured by PCR on days 0,7 and 14. A baseline fecal and oropharyngeal sample will be obtained on Day 0 prior to starting dosing of drugs.
  Other Names: Telehealth monitoring
  Arms: Fluvoxamine Arm
Combination Product: Fluvoxamine, Bromhexine — The subjects received fluvoxamine (immediate release) 50 mg, 1 tablet in the morning and 50 mg 2 tablets before bedtime, orally after meals. For a total of 14 days, the first two days and the last two days, 50 mg 1 tablet in the morning and 50 mg 1 tablet at bedtime. Co- administration with bromhexine 8 mg, 1 tablet twice taken after meals and taken at least 8 hours apart, for 10 days.
  All enrolled patients will be provided a thermometer as well as a fingertip probe pulse oximeter, with the specific instructions to monitor both temperature at oxygen saturation at the time of daily oral administration of drug. In addition, Oropharyngeal swab samples will be collected for viral shedding as measured by PCR on days 0, 7 and 14. Fecal and blood samples will be collected for viral shedding as measured by PCR on days 0,7 and 14. A baseline fecal and oropharyngeal sample will be obtained on Day 0 prior to starting dosing of drugs.
  Other Names: Telehealth monitoring
  Arms: Fluvoxamine in Combination with Bromhexine Arm
Combination Product: Fluvoxamine, Cyproheptadine — The subjects received fluvoxamine (immediate release) 50 mg, 1 tablet in the morning and 50 mg 2 tablets before bedtime, orally after meals. For a total of 14 days, the first two days and the last two days, 50 mg 1 tablet in the morning and 50 mg 1 tablet at bedtime. Co- administration with cyproheptadine 4 mg, 1 tablet, three times, orally after meals and should be taken every 8 hours apart, for 14 days.
  All enrolled patients will be provided a thermometer as well as a fingertip probe pulse oximeter, with the specific instructions to monitor both temperature at oxygen saturation at the time of daily oral administration of drug. In addition, Oropharyngeal swab samples will be collected for viral shedding as measured by PCR on days 0, 7 and 14. Fecal and blood samples will be collected for viral shedding as measured by PCR on days 0,7 and 14. A baseline fecal and oropharyngeal sample will be obtained on Day 0 prior to starting dosing of drugs.
  Other Names: Telehealth monitoring
  Arms: Fluvoxamine in Combination with Cyproheptadine Arm
Drug: Niclosamide Pill — The subjects received 1 tablet of niclosamide 1000 mg orally in divided doses twice a day. After meals in the morning and evening for a total of 14 days.
  All enrolled patients will be provided a thermometer as well as a fingertip probe pulse oximeter, with the specific instructions to monitor both temperature at oxygen saturation at the time of daily oral administration of drug. In addition, Oropharyngeal swab samples will be collected for viral shedding as measured by PCR on days 0, 7 and 14. Fecal and blood samples will be collected for viral shedding as measured by PCR on days 0,7 and 14. A baseline fecal and oropharyngeal sample will be obtained on Day 0 prior to starting dosing of drugs.
  Other Names: Telehealth monitoring
  Arms: Niclosamide Arm
Combination Product: Niclosamide, Bromhexine — The subjects received 1 tablet of niclosamide 1000 mg orally in divided doses twice a day. After meals in the morning and evening for a total of 14 days. Co-administration with bromhexine 8 mg, 1 tablet twice taken after meals and taken at least 8 hours apart, for 10 days.
  All enrolled patients will be provided a thermometer as well as a fingertip probe pulse oximeter, with the specific instructions to monitor both temperature at oxygen saturation at the time of daily oral administration of drug. In addition, Oropharyngeal swab samples will be collected for viral shedding as measured by PCR on days 0, 7 and 14. Fecal and blood samples will be collected for viral shedding as measured by PCR on days 0,7 and 14. A baseline fecal and oropharyngeal sample will be obtained on Day 0 prior to starting dosing of drugs.
  Other Names: Telehealth monitoring
  Arms: Niclosamide in Combination with Bromhexine Arm

SUMMARY:
There is an urgent need to identify effective treatments for SARS-CoV-2 infection that helps people recover quicker and reduces the need for hospital admission. The investigators develop an open, adaptive, platform trial to evaluate treatments, Fluvoxamine, Bromhexine, Cyproheptadine, and Niclosamide suitable for use in the community for treating COVID-like-illness that might help people recover sooner and prevent hospitalisation.

DETAILED DESCRIPTION:
There is an urgent need to identify interventions against COVID-19 suitable for wide use in the community that have been proven to be effective in reducing symptom duration or hospitalisation. There is urgent need to know whether potential COVID-19 treatments such as Fluvoxamine, Bromhexine, Cyproheptadine, and Niclosamide that are available for rapid pragmatic evaluation might modify the course of COVID-19 infections, particularly among those who are at higher risk of complications, such as those aged 50 years and over with comorbidity and those aged 65 years and over.

Most reported trials have been conducted in hospital settings, and there is little evidence from community settings, where most people with COVID-19 receive care and where deployment of effective early treatment could speed time to recovery and reduce complications. The investigators established a multi-arm, adaptive platform, randomised controlled trial for community treatment of COVID-19 syndromic illness in people at higher risk of an adverse illness course.

ELIGIBILITY:
Inclusion Criteria:

* COVID-1 9 patients with mild symptoms and the results were confirmed by Antigen Test Kit or PCR for SARS-CoV-2.
* People who have symptoms consistent with COVID-19 and test positive for SARS-CoV-2 infection within 48 hours of being known.
* Participants are 18 years of age or older.

Exclusion Criteria:

* Almost recovered (generally much improved and symptoms now mild or almost absent)
* Judgement of the recruiting clinician deems ineligible.
* Previous randomisation to an arm of the trial
* Pregnancy
* Breastfeeding
* Known severe hepatic impairment.
* Known severe renal impairment.
* Currently taking Fluvoxamine, Bromhexine, Cyproheptadine, or Niclosamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Hospital admission or mortality related to COVID-19 | Within 28 days
  Contacts with health services reported by patients and/or captured by reports of patients' medical records
Time taken to self- report recovery | Enrolment through final day of participation
  Patient reports the day they feel recovered
Progression to severe COVID-19 Disease | Enrolment through final day of participation
  O2 saturation <92% on room air (in two consecutive measurements at least 2 hours apart) OR 2) requirement of hospitalization OR 3) need for artificial ventilation OR 4) death.

SECONDARY OUTCOMES:
Reduction (change) in GI viral shedding (by PCR) | Days 0,7,14
  Fecal swabs
Change in respiratory viral clearance (by PCR) | Days 0,7,14
  Oropharyngeal swabs
Time to resolution of a fever | Enrolment through final day of participation
  Online diary
Negative effects on well being | Days 0,7,15,28,60
  WHO 5 Well Being Index via online diary or telephone

OTHER OUTCOMES:
Incidence of Adverse Events (AEs) | Enrolment through 30 days after final day of participation
  Composite counts by Adverse Events and Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Dhammika Leshan Wannigama, MD PhD, Principal Investigator — Chulalongkorn University; Cameron Hurst, PhD, Study Chair — QIMR Berghofer Medical Research Institute; Kanokpoj Chanpiwat, MD, Study Chair — Rajvithi Hospital; Shuichi Abe, MD, Study Chair — Yamagata Prefectural Central Hospital; Katika Akksilp, MD, Study Director — Ministry of Health, Thailand
Locations (3):
- Thailand (3):
  - Rajvithi Hospital, Ratchathewi, Bangkok
  - Vibhavadi Hospital, Bangkok
  - Chiangmai Neurological Hospital, Chiang Mai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wannigama DL, Hurst C, Phattharapornjaroen P, Hongsing P, Sirichumroonwit N, Chanpiwat K, Rad S M AH, Storer RJ, Ounjai P, Kanthawee P, Ngamwongsatit N, Kupwiwat R, Kupwiwat C, Brimson JM, Devanga Ragupathi NK, Charuluxananan S, Leelahavanichkul A, Kanjanabuch T, Higgins PG, Badavath VN, Amarasiri M, Verhasselt V, Kicic A, Chatsuwan T, Pirzada K, Jalali F, Reiersen AM, Abe S, Ishikawa H; COVID-EarlyMed Trial Team. Early treatment with fluvoxamine, bromhexine, cyproheptadine, and niclosamide to prevent clinical deterioration in patients with symptomatic COVID-19: a randomized clinical trial. EClinicalMedicine. 2024 Mar 14;70:102517. doi: 10.1016/j.eclinm.2024.102517. eCollection 2024 Apr. PMID 38516100